CLINICAL TRIAL: NCT05281679
Title: The Effects of Blood Flow Restriction With Low-intensity Resistance Training Versus Traditional Resistance Exercise on Lower Limb Strength, Walking Capacity, and Balance in Patients With Ischemic Stroke: (BFR-Stroke RESILIENCE Trial)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ishtiaq Ahmed, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-13022260-199-207631
Record Dates: First submitted 2022-02-17; First posted 2022-03-16 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Stroke, Ischemic; Cerebrovascular Accident
Keywords: Blood flow restriction; Resistance exercise; Mobility; Walking capacity
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-intensity resistance exercise with blood flow restriction group (L-BFR). (Experimental): All the participants in the low-intensity resistance exercise with blood flow restriction group (L-BFR) will receive 3 sessions of low-intensity resistance training with blood flow restriction for a total of 5 weeks.
  Interventions: Other: Low-intensity resistance exercise with blood flow restriction group (L-BFR)
- High-intensity resistance exercise without blood flow restriction group (H-BFR). (Active Comparator): All the participants in the high-intensity resistance exercise without blood flow restriction group (H-BFR) will receive 3 sessions of high-intensity resistance training without blood flow restriction for a total of 5 weeks.
  Interventions: Other: High-intensity resistance exercise without blood flow restriction group (H-BFR).

INTERVENTIONS:
Other: Low-intensity resistance exercise with blood flow restriction group (L-BFR) — The blood flow restriction training group will perform 3 sets of Sandbag (SB) resistance exercises, targeting the large muscles of the legs, at 40% of 1-RM. The SB protocol consists of 3 sets of 4 SB exercises. Each set consists of 10 repetitions of 1-RM with a 1-min recovery interval between sets and 3-min between exercises. Blood flow to the active muscle during training will be restricted by a blood flow restriction band (tourniquet) placed at the proximal end of the lower limbs. When the subjects performed training with BFR, the proximal portions of their lower limbs will be compressed at the pressure of 120-160 mmHg by electronically controlled air pressure belts. The air pressure belt will be inflated before the exercise and will remain inflated during one-minute intervals between the sets and will be deflated during the three-minute interval between the exercise.
  Arms: Low-intensity resistance exercise with blood flow restriction group (L-BFR).
Other: High-intensity resistance exercise without blood flow restriction group (H-BFR). — The high-intensity restriction training group will perform 3 sets of Sandbag (SB) resistance exercises, targeting the large muscles of the legs, at 80% of 1-RM. The SB protocol consist of 3 sets of 4 SB exercises. Each set consists of 10 repetitions of 1-RM with a 1-min rest interval between sets and 3-min between exercises.
  Arms: High-intensity resistance exercise without blood flow restriction group (H-BFR).

SUMMARY:
Stroke is the leading neurological disease in the world that causes long-term disability. The most common cause of disability after stroke is motor impairment resulting from brain damage which ultimately causes mobility and functional limitation. Worldwide, the incidence of stroke has been increased by 30% in the last decade. In Europe, more than one million cases have been reported each year and six million stroke survivors are known to be alive till now. The annual estimated cause of stroke treatment in Europe is twenty-seven billion Euros. By 2030, it is estimated that the cost of stroke treatment will be triple the current amount and can reach up to 184 billion dollars. Therefore, it is necessary to develop an economical rehabilitation program that prevents or reduces long-term disability after stroke.

DETAILED DESCRIPTION:
Blood flow restriction combined with resistance training may be an economic and time-efficient alternative to High-Intensity Training to manage the risk factors of stroke and can also be useful in reducing stroke-related impairment effectively. During BFRT, the blood flow of the exercising muscle is restricted by placing the inflated tourniquets at the most proximal part of the legs or arms. By restricting the blood flow to the limbs, the desired muscle group will work in an ischemic environment and can trigger a significant increase in muscle mass, power, and strength by recruiting the fast-twitch muscle fibers. BFRT could be a promising type of exercise for high-risk groups of patients such as Cardiovascular disease, stroke, etc, and the hypertrophy responses induced by is comparable to that produced by high-intensity training. It was found that BFRT and high-intensity training produced similar effects on both systolic, diastolic blood pressure, and heart rate (HR) in young individuals and older adults. Previous evidence from neurological studies showed that resistance combined with blood flow restriction can improve muscle strength, balance, walking capacity, and cognitive function in Multiple Sclerosis and spinal cord injury patients. Recent study showed that BFR combined with resistance training has improved brain-derived neurotrophic factor (BDNF) and vascular endothelial growth factor (VEGF) and rate of perceived exertion in ischemic stroke patients. Kaatsu training society also reported a few cases in which BFRT has produced a positive effect on the recovery of stroke patients, but the evidence is insufficient to support this assertion.

ELIGIBILITY:
Inclusion Criteria:

* All the participants will be evaluated to be in stable Cardio-vascular condition i,e ACSM Class B.
* 18 to 90 years of age.
* More than 1 month of stroke onset.
* First ever unilateral ischemic stroke.
* Being able to walk 10 m independently with or without an assistive device.
* Being an independent ambulator (Functional Ambulation Scale>3).
* Muscle tension of the modified Ashworth scale was lower than grade.

Exclusion Criteria

* People with a history of mental illness.
* People with obvious cognitive impairments.
* Combination with peripheral neuropathy.
* Having resting blood pressure above 160/100 mmHg even after taking medications.
* Hemorrhagic stroke
* Cardiovascular comorbidity (aortic stenosis, depression of ST-segment, heart failure, arrhythmias, unstable angina, hypertrophic cardiomyopathy).
* Transient ischemic attack.
* By-pass surgery in the recent three months
* Any 0ther musculoskeletal problems that prevented the participants from doing resistance training
* People who have taken antipyretics, analgesics, dopamine, and other drugs that affect autonomic nerve function within 2 weeks.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-03-20 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Change score of Sit to stand Test | Baseline, Post-intervention (Approximately 5 weeks), follow-up (up to 3 Months)
  Five time sit to stand test will be used to assess lower extremity muscle strength, balance and risk of fall in stroke patients. The test measure amount of time taken to complete five repetitions of sit to stand task. The test will be performed with standard height chair without an armrest and with straight back (43-45 cm high). He patients will be instructed to stand up and sit down as quickly as possible 5 times, keeping their arms folded across their chest. Timing began when the patient's back left the backrest and stopped once the back touched the backrest for the fifth time.
Change score of 10 Meter walk Test | Baseline, Post-intervention (Approximately 5 weeks)
  The Comfortable 10-m Walk Test (10 MWT) will be used to determine the speed of comfortable walking. The test will be applied in a 14-m corridor. The patients will be instructed to walk comfortably and allowed to use walking aid. At the 2nd meter, the stopwatch will be started and stopped when the patient reached the 12th meter. Walking time and number of steps will be assessed to calculate gait speed (m/s), stride length (m), and cadence (steps/min). After three trials, the average of the three trials will be recorded as m/s.
Change score of Timed up and Go Test (TUG) | Baseline, Post-intervention (Approximately 5 weeks)
  The Timed Up & Go test is a functional mobility test used to assess dynamic balance, transfer, and gait. The patient is instructed to stand up from a chair (46 cm high) with support for the arms, walk for a short distance (3 m), turn, go back and sit down as quickly as possible. The stopwatch will be used to measure the time to perform these tasks from start to end. The patients will be allowed to use their walking aids. After three trials, the average of the three trials will be recorded.
Change score of 6 Minute walk Test | Baseline, Post-intervention (Approximately 5 weeks)
  The walking distance will be measured by the 6 Minute walk Test (6MWT), the most commonly used for measuring the physical performance of individuals after stroke. The patients will be asked to walk as far as possible throughout the 30-meter course within 6 minutes by following the standardized instructions provided by the physiotherapist. Participants will be allowed by the physiotherapist to use aiding device if necessary. Physiotherapist will guard the participants during the walk test but will not offer any assistance or support to the participant.
Change score of Barthel Index | Baseline, Post-intervention (Approximately 5 weeks)
  The Barthel Index measures a person's performance in activities of daily living. The Barthel Index consists of 10 items of mobility and self care activities of daily living. This score will be measured on admission and at the end of intervention (at the end of 5th week). The minimum score is 0 and the maximum is 100. A higher score indicates a better outcome.

SECONDARY OUTCOMES:
Change score of Hospital Anxiety and Depression Scale (HADS) | Baseline, Post-intervention (Approximately 5 weeks)
  The Hospital Anxiety and Depression Scale (HADS) is a fourteen-item scale scoring from 0 to 3 for each item. The first seven items relate to anxiety (HADS-A), and the remaining seven items relate to depression (HADS-D). The global scoring ranges from 0 to 42 with a cut-off point of 8/21 for anxiety and 8/21 for depression. The higher the score, the greater anxiety or depression symptoms. HADS will be performed at the beginning and after four weeks of treatment.
Attendance | Number of sessions attended will be measured during the 5 weeks of intervention protocol.
  Attendance of training sessions measured via Hospital entry sheet.
Adverse Events | Any adverse event reported during the 5 weeks of intervention protocol.
  Any adverse event or near miss is required to be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Rustem Mustafaoglu, PhD, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Göztepe Prof. Dr. Süleyman Yalçın City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Freitas EDS, Miller RM, Heishman AD, Aniceto RR, Larson R, Pereira HM, Bemben D, Bemben MG. The perceptual responses of individuals with multiple sclerosis to blood flow restriction versus traditional resistance exercise. Physiol Behav. 2021 Feb 1;229:113219. doi: 10.1016/j.physbeh.2020.113219. Epub 2020 Oct 24. PMID 33250152
- [Result] Du X, Chen W, Zhan N, Bian X, Yu W. The effects of low-intensity resistance training with or without blood flow restriction on serum BDNF, VEGF and perception in patients with post-stroke depression. Neuro Endocrinol Lett. 2021 Aug 28;42(4):229-235. PMID 34436843
- [Derived] Ahmed I, Mustafaoglu R, Erhan B. The effects of low-intensity resistance training with blood flow restriction versus traditional resistance exercise on lower extremity muscle strength and motor functionin ischemic stroke survivors: a randomized controlled trial. Top Stroke Rehabil. 2024 May;31(4):418-429. doi: 10.1080/10749357.2023.2259170. Epub 2023 Sep 19. PMID 37724785